CLINICAL TRIAL: NCT00107263
Title: A Randomized, Controlled, Open-Label Trial of Empiric Prophylactic vs. Delayed Use of Zoledronic Acid for Prevention of Bone Loss in Postmenopausal Women With Breast Cancer Initiating Therapy With Letrozole After Tamoxifen
Brief Title: Zoledronate in Preventing Bone Loss in Postmenopausal Women Who Are Receiving Letrozole for Stage I, Stage II, or Stage IIIA Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NCCTG-N03CC; CDR0000413877 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer; Osteoporosis
Keywords: osteoporosis; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms; Osteoporosis | interventions — Letrozole; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: letrozole + zoledronate (Experimental): Patients receive oral letrozole once daily. Patients also receive zoledronate IV over 15 minutes once every 6 months.
  Treatment continues for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: letrozole; Drug: zoledronic acid
- Arm II: letrozole + zoledronate (Experimental): Patients receive oral letrozole once daily. Patients with radiologic evidence of bone loss after 1 year of letrozole therapy receive zoledronate as in arm I.
  Treatment continues for up to 5 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: letrozole; Drug: zoledronic acid

INTERVENTIONS:
Drug: letrozole
Drug: zoledronic acid

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by lowering the amount of estrogen the body makes. Zoledronate may prevent bone loss in patients who are receiving letrozole. It is not yet known which schedule of zoledronate is more effective in preventing bone loss in patients with breast cancer.

PURPOSE: This randomized phase III trial is studying two different schedules of zoledronate to compare how well they work in preventing bone loss in postmenopausal women who are receiving letrozole for stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness of zoledronate vs standard care in reducing bone loss during the first 12 months of study treatment in postmenopausal women with stage I-IIIA breast cancer initiating letrozole after prior treatment with tamoxifen.
* Compare the effect of immediate vs delayed zoledronate, annually at 2-5 years post-baseline, in reducing bone loss in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are stratified according to duration of prior tamoxifen therapy (≤ 2 years vs > 2 years); time since tamoxifen therapy was discontinued (< 1 vs ≥ 1 year); prior adjuvant chemotherapy (yes vs no); and baseline total lumbar spine or femoral neck bone mineral density (BMD) T-score (> -1 standard deviation [SD] vs between -1 to -2 SD). Patients are randomized to 1 of 2 treatment arms.

* Arm I (immediate therapy): Patients receive oral letrozole once daily. Patients also receive zoledronate IV over 15 minutes once every 6 months.
* Arm II (delayed therapy): Patients receive oral letrozole as in arm I. Patients with radiologic evidence of bone loss after 1 year of letrozole therapy receive zoledronate as in arm I.

In both arms, treatment continues for up to 5 years in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 550 patients (275 per treatment arm) will be accrued for this study within 28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Stage I, II, or IIIA disease
* Completed ≤ 6 years of adjuvant tamoxifen therapy
* Total baseline lumbar spine or femoral neck bone mineral density T-score below -2.0 standard deviation (e.g., a patient with a T-score of -2.1 in ineligible; a patient with a T-score of -1.9 is eligible)
* No clinical or radiological evidence of recurrent or metastatic disease
* Hormone receptor status:

  * Estrogen receptor- and/or progesterone receptor-positive

PATIENT CHARACTERISTICS:

Age

* Postmenopausal

Sex

* Female

Menopausal status

* Postmenopausal, defined by 1 of the following:

  * Over 55 years of age with cessation of menses
  * 55 years of age and under with spontaneous cessation of menses for > 1 year
  * 55 years of age and under with spontaneous cessation of menses for ≤ 1 year, but amenorrheic (e.g., spontaneous or secondary to hysterectomy) with postmenopausal estradiol levels (< 5 ng/dL)
  * Undergone bilateral oophorectomy

Performance status

* ECOG 0-2

Life expectancy

* At least 5 years

Hematopoietic

* WBC ≥ 3,000/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* AST ≤ 3 times ULN

Renal

* Creatinine < 2.0 mg/dL
* No hypercalcemia (i.e., calcium > 1 mg/dL above ULN within the past 6 months)
* No hypocalcemia (i.e., calcium > 0.5 mg/dL below lower limit of normal within the past 6 months)

Other

* No uncontrolled infection
* No uncontrolled diabetes mellitus
* No uncontrolled thyroid dysfunction
* No disease affecting bone metabolism (e.g., hyperparathyroidism, hypercortisolism, Paget's disease, or osteogenesis imperfecta)
* No malabsorption syndrome
* No uncontrolled seizure disorder associated with falls
* No known hypersensitivity to zoledronate or other bisphosphonates, letrozole, calcium, or cholecalciferol (vitamin D)
* No mental illness that would preclude giving informed consent
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No other non-malignant systemic disease
* No clinical or radiologic evidence of existing fracture in the lumbar spine and/or total hip
* No history of fracture with low intensity or not associated with trauma
* No contraindication to spinal dual energy x-ray absorptiometry (DEXA) due to any of the following:

  * History of surgery at the lumbosacral spine, with or without implantable devices
  * Scoliosis with a Cobb angle > 15° at the lumbar spine
  * Immobility, hyperostosis, or sclerotic changes at the lumbar spine
  * Evidence of sufficient sclerotic abdominal aorta that would interfere with DEXA scan
  * Any disease of the spine that would preclude proper acquisition of a lumbar spine DEXA
* Considered reliable

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* Prior parathyroid hormone allowed provided it was not administered for > 1 week
* More than 6 months since prior anabolic steroids or growth hormone
* More than 12 months since prior endocrine therapy (including estrogen) except for the following:

  * Tamoxifen
  * Insulin
  * Oral hypoglycemics
  * Thyroid hormone
  * Steroid inhalers
* More than 12 months since prior systemic corticosteroids except short-term corticosteroids to prevent or treat chemotherapy-induced nausea and vomiting or acute respiratory illness

  * Concurrent short-term corticosteroids allowed
* No other concurrent hormonal therapy
* No concurrent parathyroid hormone

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Prior systemic sodium fluoride allowed provided it was not administered for > 3 months within the past 2 years
* More than 3 weeks since prior oral bisphosphonates
* More than 2 weeks since prior and no concurrent drugs known to affect the skeleton (e.g., calcitonin, mithramycin, or gallium nitrate)
* More than 30 days since prior systemic investigational drugs and/or devices
* More than 7 days since prior topical investigational drugs
* No prior IV bisphosphonates
* No prior aromatase inhibitor therapy
* No concurrent calcitonin, sodium fluoride, or Tibolone
* No other concurrent anticancer therapy
* No other concurrent bisphosphonates
* No other concurrent investigational drugs or devices

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Average intra-patient change in total lumbar spine (L1-L4) bone mineral density (BMD) as measured by dual energy x-ray absorptiometry at baseline and 1 year after completion of study treatment | at 12 months

SECONDARY OUTCOMES:
BMD (lumbar spine) annually for 5 years after completion of study treatment | Up to 5 years
Incidence of osteoporosis | Up to 5 years
Loss of bone density | Up to 5 years
Incidence of bone fractures | Up to 5 years
Time to disease progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Hines, MD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] Hines SL, Mincey B, Dentchev T, Sloan JA, Perez EA, Johnson DB, Schaefer PL, Alberts S, Liu H, Kahanic S, Mazurczak MA, Nikcevich DA, Loprinzi CL. Immediate versus delayed zoledronic acid for prevention of bone loss in postmenopausal women with breast cancer starting letrozole after tamoxifen-N03CC. Breast Cancer Res Treat. 2009 Oct;117(3):603-9. doi: 10.1007/s10549-009-0332-2. Epub 2009 Feb 12. PMID 19214743
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716